CLINICAL TRIAL: NCT05575037
Title: Mechanisms of Benefit of IL4RA Inhibition in Aspirin-Exacerbated Respiratory Disease: MARINER
Brief Title: Mechanisms of Benefit of IL4RA Inhibition in Aspirin-Exacerbated Respiratory Disease
Acronym: MARINER
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Tanya Laidlaw, MD, Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022P002407; U19AI095219 (NIH)
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Nasal Polyps; Asthma, Aspirin-Induced; Aspirin-Exacerbated Respiratory Disease; Aspirin-Sensitive Asthma With Nasal Polyps
MeSH Terms: conditions — Nasal Polyps; Asthma, Aspirin-Induced | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dupilumab (Experimental): Subjects will receive dupilumab (300mg every-other-week for 8 weeks).
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — 8-week trial of dupilumab (an anti-IL-4a) in patients with AERD.
  Other Names: Dupilumab Prefilled Syringe [Dupixent]

SUMMARY:
The overall aim of the study is to determine the clinical efficacy and mechanisms of action of anti-IL-4a (dupilumab) as treatment for patients with Chronic Rhinosinusitis with Nasal Polyposis (CRSwNP) and Aspirin-Exacerbated Respiratory Disease (AERD).

DETAILED DESCRIPTION:
The protocol involves an 8-week study of dupilumab in patients with CRSwNP and/or AERD. Participants will have 4 total doses of dupilumab administered, with each dose administered every 2 weeks. There will be full clinical assessments and biospecimen collections at Baseline (Visit 1), Week 2 (Visit 2), and Week 8 (Visit 3).

ELIGIBILITY:
Key Inclusion Criteria:

1. History of AERD, defined as meeting the diagnostic triad with:

   1. History of physician-diagnosed asthma and
   2. History of physician-diagnosed nasal polyposis and
   3. History of pathognomonic reactions to aspirin or other nonselective COX inhibitors.
2. Visible nasal polyps bilaterally on otoscope physical exam at the time of screening.
3. Evidence of sense of smell impairment, with a University of Pennsylvania Smell Identification Test (UPSIT) score of <34.
4. Stable asthma (no glucocorticoid burst for at least 4 weeks prior to Visit 1, and no hospitalizations or ER visits for asthma for at least the prior 3 months).
5. Consistent (daily) use of an intranasal steroid for at least 4 weeks prior to Screening.
6. No current smoking (not more than one instance of smoking in the last 3 months).
7. For females: Practicing FDA-approved methods of birth control for the duration of the study. Female participants of childbearing potential must have a negative pregnancy test upon study entry.

Key Exclusion Criteria:

1. Use of investigational drugs within 12 weeks of Screening.
2. Use of any biologic agent within 4 months prior to Screening.
3. Use of systemic (enteral or injected) glucocorticoids within 4 weeks prior to Screening.
4. History of any sinonasal surgery within 4 months prior to Screening
5. Current use of zileuton
6. Current use of high-dose aspirin therapy (no more than 325 mg aspirin per day will be allowed)
7. Pregnant, nursing, or planning to become pregnant

Note: Other inclusion and exclusion criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Nasal fluid levels of LTE4 | At Week 8 (Visit 3)
  The nasal fluid levels of LTE4 will be measured at week 8 and will serve as a surrogate biomarker of respiratory mast cell activation or burden.

SECONDARY OUTCOMES:
Nasal fluid levels of albumin | At Week 8 (Visit 3)
  The nasal fluid levels of albumin will be measured at week 8 and serve as a surrogate biomarker of nasal epithelial cell integrity.
Sense of smell - University of Pennsylvania Smell Identification Test (UPSIT) | At Week 8 (Visit 3)
  Patients' sense of smell will be assessed at week 8 using the UPSIT. The UPSIT scale goes from 0 to 40, with 0 being worse (no scents identified) and 40 being best (all scents identified)
Rhinoscopic Total Polyp Score (TPS) | At Week 8 (Visit 3)
  The extent of patients' nasal polyps will be assessed at week 8 using a TPS. The TPS scale goes from 0 (no polyps) to 8 (large polyps bilaterally), with 0 being best and 8 being worst.
Peak Nasal Inspiratory Flow (PNIF) | At Week 8 (Visit 3)
  Patients' nasal congestion will be assessed at week 8 by a PNIF. PNIF goes from 0 mL (no airflow) to 500 mL of airflow, with 0 being worst.
Quality of life - 22-Item Sino-Nasal Outcome Test (SNOT-22) | At Week 8 (Visit 3)
  Quality of life will be assessed at week 8 with a SNOT-22. For the SNOT-22, the scores range from 0 (no symptoms, excellent disease control) to 110 (maximum sinus symptoms, poor disease control).
Lung function - Forced Expiratory Volume 1 (FEV1) | At Week 8 (Visit 3)
  Patients' lung function will be assessed at week 8 with an FEV1.
Asthma control - Asthma Control Questionnaire-6 (ACQ-6) | At Week 8 (Visit 3)
  Asthma control will be measured at week 8 with an ACQ-6. For the ACQ-6, scores ranging from 0 (well-controlled) to 6 (extremely poorly-controlled). A lower score indicates better asthma control.
Number of treatment-related adverse events (AEs) and serious adverse events (SAEs) leading to study drug discontinuation | At Week 8 (Visit 3)
  Safety will be measured by the number of treatment-related AEs and SAEs leading to dupilumab discontinuation.

OTHER OUTCOMES:
Change in sense of smell - University of Pennsylvania Smell Identification Test (UPSIT) | 2 weeks (between Visit 1 and Visit 2) and 8 weeks (between Visit 1 and Visit 3)
  Change from Visit 1 to Visit 2 and from Visit 1 to Visit 3 in UPSIT. The UPSIT scale goes from 0 to 40, with 0 being worse (no scents identified) and 40 being best (all scents identified)
Change in Rhinoscopic Total Polyp Score (TPS) | 2 weeks (between Visit 1 and Visit 2) and 8 weeks (between Visit 1 and Visit 3)
  Change from Visit 1 to Visit 2 and from Visit 1 to Visit 3 in TPS. The TPS scale goes from 0 (no polyps) to 8 (large polyps bilaterally), with 0 being best and 8 being worst.
Change in Peak Nasal Inspiratory Flow (PNIF) | 2 weeks (between Visit 1 and Visit 2) and 8 weeks (between Visit 1 and Visit 3)
  Change from Visit 1 to Visit 2 and from Visit 1 to Visit 3 in PNIF. PNIF goes from 0 mL (no airflow) to 500 mL of airflow, with 0 being worst.
Change in 22-Item Sino-Nasal Outcome Test (SNOT-22) | 2 weeks (between Visit 1 and Visit 2) and 8 weeks (between Visit 1 and Visit 3)
  Change from Visit 1 to Visit 2 and from Visit 1 to Visit 3 in SNOT-22. For the SNOT-22, the scores range from 0 (no symptoms, excellent disease control) to 110 (maximum sinus symptoms, poor disease control).
Change in lung function - Forced Expiratory Volume 1 (FEV1) | 2 weeks (between Visit 1 and Visit 2) and 8 weeks (between Visit 1 and Visit 3)
  Change from Visit 1 to Visit 2 and from Visit 1 to Visit 3 in FEV1.
Change in Asthma control - Asthma Control Questionnaire-6 (ACQ-6) | 2 weeks (between Visit 1 and Visit 2) and 8 weeks (between Visit 1 and Visit 3)
  Change from Visit 1 to Visit 2 and from Visit 1 to Visit 3 in ACQ-6. For the ACQ-6, scores ranging from 0 (well-controlled) to 6 (extremely poorly-controlled). A lower score indicates better asthma control.
Change in Nasal fluid levels of eicosanoids | weeks (between Visit 1 and Visit 2) and 8 weeks (between Visit 1 and Visit 3)
  Change from Visit 1 to Visit 2 and from Visit 1 to Visit 3 in nasal fluid eicosanoid levels.
Change in Nasal fluid levels of albumin | 2 weeks (between Visit 1 and Visit 2) and 8 weeks (between Visit 1 and Visit 3)
  Change from Visit 1 to Visit 2 and from Visit 1 to Visit 3 in nasal fluid albumin levels.
Change in urinary levels of eicosanoids | 2 weeks (between Visit 1 and Visit 2) and 8 weeks (between Visit 1 and Visit 3)
  Change from Visit 1 to Visit 2 and from Visit 1 to Visit 3 in urinary eicosanoid levels.
Change in serum tryptase | 2 weeks (between Visit 1 and Visit 2) and 8 weeks (between Visit 1 and Visit 3)
  Change from Visit 1 to Visit 2 and from Visit 1 to Visit 3 in serum tryptase levels.
Change in IgE levels | 2 weeks (between Visit 1 and Visit 2) and 8 weeks (between Visit 1 and Visit 3)
  Change from Visit 1 to Visit 2 and from Visit 1 to Visit 3 in nasal fluid and plasma levels of IgE.
Change in eosinophilic cationic protein (ECP) | 2 weeks (between Visit 1 and Visit 2) and 8 weeks (between Visit 1 and Visit 3)
  Change from Visit 1 to Visit 2 and from Visit 1 to Visit 3 in nasal fluid levels of ECP.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya M Laidlaw, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-11): https://cdn.clinicaltrials.gov/large-docs/37/NCT05575037/Prot_SAP_000.pdf